CLINICAL TRIAL: NCT06875050
Title: Effect of Antioxidant Supplements on Oxidative Stress, Disease Severity and Bacterial Infection in Cystic Fibrosis Children
Brief Title: Antioxidant Supplements in Cystic Fibrosis Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, Lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MS 98/2024
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1(Extra care group) (Experimental)
  Interventions: Other: Mediterranean diet; Dietary Supplement: Antioxidant Supplement
- Arm 2 (Active Comparator)
  Interventions: Other: Mediterranean diet; Dietary Supplement: Fat soluble vitamins supplementation

INTERVENTIONS:
Other: Mediterranean diet — Tailored dietary plan following Mediterranean diet to cover macronutrients needs according to recommended daily allowance (RDA) for age
Dietary Supplement: Fat soluble vitamins supplementation — Fat soluble vitamins supplementation (150 μg vitamin A, 2000 IU vitamin D, 100 mg vitamin E and 1000 μg vitamin K).
  Arms: Arm 2
Dietary Supplement: Antioxidant Supplement — Antioxidant supplements in specific doses in oral liquid form (200 mg vitamin E, 300 mg vitamin C, 90 μg Se, 500 μg vitamin A, 30 mg zinc, 3 mg copper and 2000 IU vitamin D).
  Arms: Arm 1(Extra care group)

SUMMARY:
This randomized controlled clinical trial included 60 pediatric patients with cystic fibrosis (CF) assigned randomly into two arms; Arm 1(extra care arm):received a tailored dietary plan following Mediterranean diet to cover macronutrients needs according to recommended daily allowance (RDA) for age, with antioxidant supplements in specific doses in oral liquid form (200 mg vitamin E, 300 mg vitamin C, 90 μg Se, 500 μg vitamin A, 30 mg zinc, 3 mg copper and 2000 IU vitamin D) for 6 months. Arm 2: recieved tailored dietary plan following Mediterranean diet as Arm 1 with fat soluble vitamins supplementation (150 μg vitamin A, 2000 IU vitamin D, 100 mg vitamin E and 1000 μg vitamin K) for 6 months. This study aimed to evaluate the effect of antioxidants supplementation on the level of oxidative stress, as measured by 3-Nitrotyrosine, bacterial colonization and diseases severity among CF children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented diagnosis of cystic fibrosis (CF) who were diagnosed according to CF Foundation guidelines based upon positive sweat tests and/or the presence of a mutation in the homozygous state or two heterozygous mutations on the gene encoding the cystic fibrosis transmembrane conductance regulator (CFTR) protein

Exclusion Criteria:

* Patients with current pulmonary exacerbations.
* Patients with severe sepsis.
* Patients with comorbid systemic illnesses.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
evaluate the effect of antioxidants supplementation on the level of oxidative stress among CF children.. | 6 months
  To evaluate the effect of antioxidants supplementation on the level of oxidative stress, as measured by 3-Nitrotyrosine, bacterial colonization and diseases severity among CF children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided